CLINICAL TRIAL: NCT04781023
Title: Evaluation of the Efficacy of an Intravaginal Treatment With Carboxymethyl-β-glucan and Polycarbophil in the Clearance of High-risk Human Papillomavirus Infection
Brief Title: Efficacy of an Intravaginal Treatment With Carboxymethyl-β-glucan and Polycarbophil in HR-HPV Clearance
Acronym: GLUCANVIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uriach Consumer Healthcare (Industry)
Collaborators: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLUCANVIR V1 15/7/2020
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilomavirus; Cervical cancer; Cervial lesions; High-Risk Papillomavirus; beta-glucans
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional, longitudinal, prospective, open label trial with a control group with randomized, consecutive recruitment for each group, to evaluate the safety and efficacy of carboxymethyl-beta-glucan and polycarbophil as a treatment for high-risk HPV infection in women without cytological alterations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Colpofix) (Experimental): intravaginal gel with carboxymtheyl beta-glucan and polycabophil
  Interventions: Device: Colpofix
- Control (No Intervention): No intervention (standard of care)

INTERVENTIONS:
Device: Colpofix — Intravaginal gel with carboxymtheyl beta-glucan and polycabophil. Posology: 1 application / day x 20 days, rest 10. Repeat 20 x 3 cycles
  Arms: Intervention (Colpofix)

SUMMARY:
These treatments are beta-glucans, polysaccharides of beta-D-glucose that, can influence the clearance of HPV infection. The objective of this study is to evaluate the efficacy of a gel with Carboxymethyl - β -Glucan and polycarbophil when applied intravaginally regarding the clearance of HPV infection.

DETAILED DESCRIPTION:
Background

Human papillomavirus (HPV) infection represents a significant source of morbidity and mortality worldwide. High-risk oncogenic HPVs cause 99.7% of cervical cancers. 80% of sexually active women will be infected with HPV at some point in their life. Most of these infections are transitory and only if they are persistent and caused by a high-risk oncogenic HPV are they an important risk factor for the development of cervical intraepithelial lesions and invasive cervical cancer. Immunity plays a key factor in eliminating HPV infection. The innate immune response constitutes the first line of defense against infection during the early stages of infection, promoting a cytokine-mediated inflammatory response which links innate immunity with the adaptive immune response. HPV evasion of these immune defense mechanisms is critical for the persistence of the infection and leads to the development of preneoplastic lesions and ultimately to cervical cancer. Through the use of adjuvant medical treatments represents a therapeutic strategy to avoid the evasion mechanisms of HPV. One of these most promising treatments is beta-glucans that seem capable of affecting the course of HPV infection.

Justification

β-glucans are a very diverse heterogeneous group of polysaccharides made up of D-glucose monomers linked by β-type glycosidic bonds.

β-glucans have been previously described in bacteria, fungi, yeasts (including brewer's yeast), plants and algae, where they play an important structural role in the cell wall or reservoir.

There are more than 6000 studies that have described the effects of glucans, mainly those of β-1,3 bonds, such as anti-inflammatory and antimicrobial properties. At least 4 receptors have been identified in mammals for the recognition of these molecules: lactosylceramide, scavengers, complement receptor 3 and dectin-1.

Commercial production of 1,3-β-glucans has been carried out by cultivating bacteria, yeasts, fungi, and plants.

Recent studies focusing on their influence on cytotoxic and helper T cells, APCs, inflammatory pathways, and oxidative burst (using reactive oxygen species to kill cells) have revealed that they may also have some anti-cancer properties. Some efforts have been made in the field of cervical cancer prevention and it has been shown that β-glucans can also affect HPV infection. Carboxymethyl β-glucan gel treatment was studied in a group of affected individuals by CIN1. This case-control study demonstrated that it has an anti-cervical cancer role in CIN1 regression. In 2010, two studies were conducted on the topic of "the influence of β-glucans" on HPV-related lesions in the genital area. "The first study found that β-glucans can treat infection-related lesions and the second study revealed the efficacy of beta-glucan treatment for HPVCIN1 lesions. These studies suggested that, in addition to the anticancer effects of beta-glucans, they also have some effects on infection by HPV, the main cause of cervical cancer.

On the other hand, the local treatment of vaginal problems has been known since ancient times, and more recently it has been favored over oral treatments due to the achievement of higher local concentrations of drugs and fewer interactions of the active principles and interference with the gastrointestinal tract. Vaginal products are marketed in the form of tablets, capsules, pessaries or ovules and semisolid forms (creams, ointments and gels), being available as products for the treatment and prevention of vaginal infections. Conventional dosage forms are associated with poor distribution and retention, primarily due to the self-cleaning action of the vagina. Among the commercialized dosage forms, semisolids, in particular gels, have been considered the preferred ones as they spread easily over the vaginal surface area. Additionally, due to their high water content, they confer moisture and lubrication effects that help alleviate the symptoms of conditions associated with vaginal dryness.

Bioadhesion refers to the binding of natural or synthetic macromolecules to a biological tissue. Mucoadhesion is considered a particular case of bioadhesion whenever the binding occurs with mucous glycoproteins (mucin) or mucous membranes. The translation of these concepts into pharmaceutical technology has been widely studied through the use of bioadhesive polymers. Among the most used in vaginal formulations are polyacrylates (such as carbomers and polycarbophils), cellulose derivatives (hydroxyethylcellulose (HEC), hydroxypropylcellulose (HPC), hydroxypropylmethylcellulose (HPMC), etc.), chitosan, hyaluronic acid and its derivatives, starch, pectin, natural gums and sodium alginate. In addition to increasing the retention time of vaginal formulations, thus promoting therapeutic duration and efficacy and improving patient comfort and adherence, these excipients also allow controlled drug release, thus improving local pharmacokinetics.

Polycarbophil and carbomer (polyacrylate) vaginal applications have been specially studied in vitro and in vivo, and have been included in various proprietary formulations as well as actual marketed products. These polymers have the additional advantage of being acidic, allowing the correction and maintenance of vaginal pH, and their acid-buffering capacity has been explored as a strategy for the treatment of bacterial vaginosis and the prevention of vaginosis recurrence for prevent the proliferation of pathogens, while promoting the restoration of the protective flora of Lactobacillus.

Polycarbophil, in particular, has been widely used for its bioadhesive properties, especially after a 1-3% polycarbophil gel was shown to maintain vaginal acidity for 3-4 days after a single application in postmenopausal women and A polycarbophil-carbomer vaginal gel was proven in women with suspected and confirmed bacterial vaginosis to show a reduction in vaginal pH in both trials, and a high clinical cure rate in confirmed vaginosis cases compared to placebo.

The objective of this study is to evaluate the efficacy of a gel with Carboxymethyl - β -Glucan and polycarbophil when applied intravaginally regarding the clearance of HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women
* between 30 and 40 years old
* HR-HPV+ test (genotypes 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68)
* normal cytology

Exclusion Criteria:

* Current or previous pregnancy ended before six weeks in relation to the start of the study.
* Vaccination against HPV.
* Clinically relevant pathology linked to immunodeficiency.
* Immunosuppressive treatment active or finished before six months in relation to the start of the study. In the specific case of corticosteroids, all women who are receiving corticosteroid treatment currently or recently (defined as the two weeks prior to the start of the study) or if she has received 2 or more cycles of corticosteroids in equal or greater than 20 mg / day of predsinone (or equivalent) orally or parenterally, for one week duration at least in the year prior to the start of the study. The use of inhaled corticosteroids, Nasal or topical are not exclusion criteria.
* Undiagnosed abnormal genital bleeding.
* Total hysterectomy.
* Presence of genital warts and other symptomatic vulvovaginal infections.
* Documented history of cervical pathology caused by HPV.
* Current systemic and / or gynecological disease that contraindicates the use of Colpofix.
* Contraindications to the use of Colpofix or known allergies to any of its components
* Simultaneous participating in a clinical study of an investigational drug or that could interfere with the use of Colpofix.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the clearance of high-risk HPV infection in women without cytological alterations upon local treatment with carboxymethyl-β-glucan and polycarbophilon the clearance of high-risk HPV infection in women without cytological alterations. | 24 months (6, 12, 18 and 24 months)
  Evaluation of the change in HPV clearance by HPV PCR test

SECONDARY OUTCOMES:
Determine the effect of local treatment with carboxymethyl - β-glucan and polycarbophil on the clearance rate of HPV | 24 months (6, 12, 18 and 24 months)
  Evaluation of HPV clearance rate by HPV PCR test
Determine the effect of local treatment with carboxymethyl - β-glucan and polycarbophil on the clearance time of HPV | 24 months (6, 12, 18 and 24 months)
  Evaluation of HPV clearance time by HPV PCR test
Change on the incidence of cytological alterations upon local treatment with carboxymethyl - β-glucan and polycarbophil during the follow-up time | 24 months (6, 12, 18 and 24 months)
  change in the incidence of cytological alterations development by cytology
Safety assessment: incidence of Adverse Events | 24 months
  Safety assessment by means of a dichotomous questionnaire and description of the adverse event, if any
Tolerance assessment: measurement of treatment acceptance by subjects | 24 months
  Tolerance acceptance by means of a dochotomous questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jesús de la Fuente Valero, MD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (1):
- Hospital Universitario Infanta Leonor, Vallecas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geller A, Shrestha R, Yan J. Yeast-Derived beta-Glucan in Cancer: Novel Uses of a Traditional Therapeutic. Int J Mol Sci. 2019 Jul 24;20(15):3618. doi: 10.3390/ijms20153618. PMID 31344853
- [Background] Chaichian S, Moazzami B, Sadoughi F, Haddad Kashani H, Zaroudi M, Asemi Z. Functional activities of beta-glucans in the prevention or treatment of cervical cancer. J Ovarian Res. 2020 Mar 5;13(1):24. doi: 10.1186/s13048-020-00626-7. PMID 32138756
- [Background] Stentella P, Biamonti A, Carraro C, Inghirami P, Mancino P, Pietrangeli D, Votano S, Lazzari P, DE Medici C. Efficacy of carboxymethyl beta-glucan in cervical intraepithelial neoplasia: a retrospective, case-control study. Minerva Ginecol. 2017 Oct;69(5):425-430. doi: 10.23736/S0026-4784.17.04053-9. PMID 28675291
- [Background] Pietrantoni E, Signore F, Berardi G, Donadio F, Donadio C. [Role of beta-glucan in the treatment of recurrent candidiasis and HPV-correlated lesions and reparative process of epidermis]. Minerva Ginecol. 2010 Feb;62(1):1-5. Italian. PMID 20186110
- [Background] Scardamaglia P, Carraro C, Mancino P, Stentella P. [Effectiveness of the treatment with beta-glucan in the HPV-CIN 1 lesions]. Minerva Ginecol. 2010 Oct;62(5):389-93. Italian. PMID 20938424
- [Background] Palmeira-de-Oliveira R, Palmeira-de-Oliveira A, Martinez-de-Oliveira J. New strategies for local treatment of vaginal infections. Adv Drug Deliv Rev. 2015 Sep 15;92:105-22. doi: 10.1016/j.addr.2015.06.008. Epub 2015 Jul 2. PMID 26144995
- [Background] Fiorilli A, Molteni B, Milani M. Successful treatment of bacterial vaginosis with a policarbophil-carbopol acidic vaginal gel: results from a randomised double-blind, placebo-controlled trial. Eur J Obstet Gynecol Reprod Biol. 2005 Jun 1;120(2):202-5. doi: 10.1016/j.ejogrb.2004.10.011. PMID 15925053